CLINICAL TRIAL: NCT07098403
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel Group Phase Ⅲ Study to Evaluate the Efficacy and Safety of SHR-1905 in Subjects With Severe Uncontrolled Asthma
Brief Title: A Trial of SHR-1905 in Subjects With Severe Uncontrolled Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1905-302
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1905 Group (Experimental)
  Interventions: Drug: SHR-1905 Injection
- SHR-1905 Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-1905 Placebo Injection

INTERVENTIONS:
Drug: SHR-1905 Injection — SHR-1905 injection.
  Arms: SHR-1905 Group
Drug: SHR-1905 Placebo Injection — SHR-1905 placebo Injection.
  Arms: SHR-1905 Placebo Group

SUMMARY:
This study is a phase III study of SHR-1905 in subjects with severe uncontrolled asthma. The purpose of the study is to evaluate efficacy and safety of SHR-1905 in subjects with severe uncontrolled asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Documented physician-diagnosed asthma for at least 12 months.
3. Participants who have received asthma controller medication with medium or high dose ICS for at least 6 months.
4. Documented treatment with a total daily dose of either medium or high dose ICS (Refer to Guidelines for the prevention and management of bronchial asthma (2024 edition)) for at least 3 months.
5. At least one additional maintenance asthma controller medication is required according to standard practice of care and must be documented for at least 3 months.
6. Pre-BD FEV1 < 80% predicted normal.
7. Objective evidence of asthma as documented.
8. Documented history of at least 2 asthma exacerbation events within 12 months, and at least one of the exacerbations should occur during the treatment of medium-to-high dose ICS.
9. ACQ-6 score ≥ 1.5 at screening and on day of baseline.
10. ePRO adherence ≥ 70% in the 7 days prior to randomization.

Exclusion Criteria:

1. Clinically significant pulmonary disease other than asthma.
2. History of cancer.
3. History of a clinically significant infection.
4. Current smokers or participants with smoking history ≥ 10 pack-yrs.
5. History of chronic alcohol or drug abuse within 12 months.
6. Hepatitis B, C or HIV.
7. Pregnant or breastfeeding.
8. History of anaphylaxis following any biologic therapy.
9. participant randomized in the current study or previous SHR-1905 studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Annual asthma exacerbation rate | During 48 weeks of treatment.

SECONDARY OUTCOMES:
Mean change from baseline in pre-dose/pre-bronchodilator (Pre-BD) forced expiratory volume in 1 Second (FEV1) | At Week 48.
Proportion of participants who had asthma exacerbations | From randomization to Week 48.
Time to the first asthma exacerbation | From randomization to Week 48.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided